CLINICAL TRIAL: NCT02932566
Title: A Randomised, Double-blind, Placebo-controlled, Phase 2 Study of the Efficacy and Safety of Pirfenidone in Patients With Heart Failure and Preserved Left Ventricular Ejection Fraction (PIROUETTE)
Brief Title: The Efficacy and Safety of Pirfenidone in Patients With Heart Failure and Preserved Left Ventricular Ejection Fraction
Acronym: PIROUETTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Manchester (Other); University of Liverpool (Other); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016CD004
Record Dates: First submitted 2016-09-27; First posted 2016-10-13 (Estimated); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Cardiac Failure
Keywords: Heart failure; Heart failure with preserved ejection fraction (HFpEF); Myocardial fibrosis; Extracellular volume fraction (ECV); Interstitial fibrosis
MeSH Terms: conditions — Heart Failure; Pulmonary Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pirfenidone (Active Comparator): Pirfenidone 801mg capsule by mouth, three times a day (target dose) for 12 months
  Interventions: Drug: Pirfenidone
- Placebo (Placebo Comparator): Placebo capsule by mouth, three times a day (target dose) for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone is an orally bioavailable, small molecule antifibrotic agent.
  Other Names: Esbriet
  Arms: Pirfenidone
Drug: Placebo — Placebo capsule, manufactured with the exact components of the Pirfenidone capsules, without the active ingredient / investigational medicinal product
  Arms: Placebo

SUMMARY:
This randomised, double-blind, placebo-controlled, phase 2 study aims to evaluate the efficacy and safety of the anti-fibrotic drug pirfenidone in the treatment of patients with heart failure and preserved left ventricular ejection fraction (HFpEF). Participants will be randomised to receive either pirfenidone or placebo, for a period of 12 months.

DETAILED DESCRIPTION:
Myocardial fibrosis is a key pathological mechanism in HFpEF. Pirfenidone is an anti-fibrotic medication licensed for the treatment of idiopathic lung fibrosis, for which it reduces lung function decline, improves progression free survival and reduces all cause mortality. In pre-clinical models, pirfenidone attenuates profibrotic pathways and is associated with regression of myocardial fibrosis. Previous studies in HFpEF populations using anti-fibrotic medications, such as angiotensin-converting enzyme (ACE) inhibitors, angiotensin-II receptor blockers and aldosterone antagonists have shown some benefit in reaching secondary end-points but do not reduce mortality. HFpEF is the final result of a number of specific underlying pathological mechanisms, and targeted treatment of these mechanisms has been cited as the future approach to further clinical trials. The investigators aim to select a population of HFpEF patients with high levels of interstitial myocardial fibrosis as measured on cardiac MRI (CMR), and randomise participants to receive pirfenidone or placebo. The primary outcome is to detect a significant reduction in myocardial fibrosis as measured on CMR after 12 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male or female; aged 40 years or older.
3. HF, defined as one symptom present at the time of screening, and one sign present at the time of screening or in the previous 12 months. Symptoms and signs are defined as:

   Symptoms: dyspnoea on exertion, orthopnoea or paroxysmal nocturnal dyspnoea Signs: peripheral oedema, crackles on chest auscultation post-cough, raised jugular venous pressure or chest x-ray demonstrating pleural effusion, pulmonary congestion, or cardiomegaly
4. Left Ventricular Ejection Fraction (LVEF) > 45% at Visit 0, (any local LVEF measurement made using echocardiography or CMR).
5. BNP ≥ 100 pg/ml or NTproBNP ≥ 300 pg/ml recorded at Visit 0. For patients in atrial fibrillation on Visit 0 ECG, BNP > 300pg/ml or NTproBNP > 900 pg/ml at Visit 0.
6. Myocardial fibrosis, defined as Extracellular Matrix (ECM) volume > 27% by CMR at Visit 0.

Exclusion Criteria:

1. Myocardial infarction, coronary artery bypass graft surgery or percutaneous coronary intervention within the previous 6 months.
2. Probable alternative cause of patient's HF symptoms that in the opinion of the investigator primarily accounts for patient's dyspnoea such as significant pulmonary disease, anaemia or obesity. Specifically, patients with the below are excluded:

   1. Severe chronic obstructive pulmonary disease (COPD) (i.e., requiring home oxygen, chronic nebuliser therapy, or chronic oral steroid therapy), or
   2. Haemoglobin < 9 g/dl, or
   3. Body mass index (BMI) > 55 kg/m2.
3. Known pericardial constriction, genetic hypertrophic cardiomyopathy, or infiltrative cardiomyopathy.
4. Clinically significant congenital heart disease.
5. Presence of severe valvular heart disease.
6. Atrial fibrillation or flutter with a resting ventricular rate > 100 bpm.
7. Any medical condition, which in the opinion of the Investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
8. Severe renal dysfunction at Visit 0, defined as estimated Glomerular Filtration Rate (eGFR) <30 mL/min (using Chronic Kidney Disease Epidemiology Collaboration Equation (CKD-EPI) calculation), or end-stage renal disease requiring dialysis.
9. History of severe hepatic impairment or liver dysfunction at Visit 0, defined as total bilirubin above the upper limit of normal (ULN) (excluding patients with Gilbert's syndrome), aspartate aminotransferase (AST) or alanine transaminase (ALT) >3 times the ULN or alkaline phosphatase >2.5 times the ULN.
10. Prolonged corrected QT interval, defined as a corrected QT interval >500 msec on ECG using Bazett formula.
11. Known hypersensitivity to any of the components of the investigational medicinal product (IMP).
12. Use of other investigational drugs at the time of enrolment, or within 30 days or 5 half-lives of enrolment, whichever is longer.
13. Fluvoxamine use within 28 days of Visit 0.
14. Contraindication to MRI scanning or gadolinium-based contrast agent
15. Pregnancy, lactation or planning pregnancy. Women of childbearing capacity are required to have a negative serum pregnancy test before treatment, must agree to pregnancy tests at study visits as defined in the Section 7.2.5 and must agree to maintain highly effective contraception during the study and for 3 months thereafter. Similarly male participants with female partners of childbearing potential must agree to maintain highly effective contraception during the study and for 3 months thereafter.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Extracellular volume fraction (ECV) | 12 months
  Absolute change in myocardial ECV, measured using CMR, from baseline to week 52

SECONDARY OUTCOMES:
Left ventricular (LV) mass | 12 months
  Absolute change in LV mass, measured using CMR, from baseline to week 52.
Left ventricular volume | 12 months
  Absolute change in LV volume, measured using CMR, from baseline to week 52.
Left ventricular ejection fraction | 12 months
  Absolute change in LV ejection fraction, measured using CMR, from baseline to week 52.
Left ventricular strain - CMR | 12 months
  Absolute change in LV strain, measured using CMR, from baseline to week 52.
Left ventricular strain - Echo | 12 months
  Absolute change in LV strain, measured using echocardiography, from baseline to week 52.
Left ventricular torsion | 12 months
  Absolute change in LV torsion, measured using echocardiography, from baseline to week 52.
Myocardial cell structure | 12 months
  Absolute change myocardial cell volume, measured using CMR, from baseline to week 52.
Diastolic function | 12 months
  Absolute change in LV diastolic function, measured using echocardiography, from baseline to week 52.
Left atrial volume | 12 months
  Absolute change in left atrial volume, measured using CMR, from baseline to week 52.
Myocardial energetic status | 12 months
  Absolute change in myocardial energetic status (Phosphocreatine (PCr) to adenosine triphosphate (ATP) ratio), measured using Phosphorus-31 Magnetic Resonance Spectroscopy (31P MRS), from baseline to week 52.
Cardiac biomarkers - N-Terminal-Pro-Brain Natriuretic Peptide (NT-Pro BNP) | 12 months
  Absolute change in NT-Pro BNP from baseline to week 13, baseline to week 26 and baseline to week 52.
Cardiac biomarkers - high-sensitivity Troponin T (hsTnT) | 12 months
  Absolute change in hsTnT from baseline to week 13, baseline to week 26 and baseline to week 52.
Patient exercise capacity | 12 months
  Absolute change in exercise tolerance, measured using 6 minute walk distance, from baseline to week 52.
Patient morbidity | 12 months
  Absolute change in health status (quality of life), HF symptoms and physical limitations, measured using change in Kansas City Cardiomyopathy Questionnaire (KCCQ) score, from baseline to week 52
All cause mortality | 12 months
  All cause mortality will be recorded but the trial is not powered for this clinical outcome
Cardiovascular mortality | 12 months
  Cardiovascular mortality will be recorded but the trial is not powered for this clinical outcome
Hospitalisation for heart failure | 12 months
  Hospitalisation for heart failure will be recorded but the trial is not powered for this clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Miller, MBChB, PhD, Principal Investigator — University of Manchester
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Taniguchi H, Ebina M, Kondoh Y, Ogura T, Azuma A, Suga M, Taguchi Y, Takahashi H, Nakata K, Sato A, Takeuchi M, Raghu G, Kudoh S, Nukiwa T; Pirfenidone Clinical Study Group in Japan. Pirfenidone in idiopathic pulmonary fibrosis. Eur Respir J. 2010 Apr;35(4):821-9. doi: 10.1183/09031936.00005209. Epub 2009 Dec 8. PMID 19996196
- [Background] King TE Jr, Bradford WZ, Castro-Bernardini S, Fagan EA, Glaspole I, Glassberg MK, Gorina E, Hopkins PM, Kardatzke D, Lancaster L, Lederer DJ, Nathan SD, Pereira CA, Sahn SA, Sussman R, Swigris JJ, Noble PW; ASCEND Study Group. A phase 3 trial of pirfenidone in patients with idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2083-92. doi: 10.1056/NEJMoa1402582. Epub 2014 May 18. PMID 24836312
- [Background] Van Erp C, Irwin NG, Hoey AJ. Long-term administration of pirfenidone improves cardiac function in mdx mice. Muscle Nerve. 2006 Sep;34(3):327-34. doi: 10.1002/mus.20590. PMID 16770778
- [Background] Yamazaki T, Yamashita N, Izumi Y, Nakamura Y, Shiota M, Hanatani A, Shimada K, Muro T, Iwao H, Yoshiyama M. The antifibrotic agent pirfenidone inhibits angiotensin II-induced cardiac hypertrophy in mice. Hypertens Res. 2012 Jan;35(1):34-40. doi: 10.1038/hr.2011.139. Epub 2011 Aug 25. PMID 21866107
- [Background] Wang Y, Wu Y, Chen J, Zhao S, Li H. Pirfenidone attenuates cardiac fibrosis in a mouse model of TAC-induced left ventricular remodeling by suppressing NLRP3 inflammasome formation. Cardiology. 2013;126(1):1-11. doi: 10.1159/000351179. Epub 2013 Jul 2. PMID 23839341
- [Derived] Lewis GA, Rosala-Hallas A, Dodd S, Schelbert EB, Williams SG, Cunnington C, McDonagh T, Miller CA. Characteristics Associated With Growth Differentiation Factor 15 in Heart Failure With Preserved Ejection Fraction and the Impact of Pirfenidone. J Am Heart Assoc. 2022 Jul 19;11(14):e024668. doi: 10.1161/JAHA.121.024668. Epub 2022 Jul 13. PMID 35861823
- [Derived] Lewis GA, Rosala-Hallas A, Dodd S, Schelbert EB, Williams SG, Cunnington C, McDonagh T, Miller CA. Impact of Myocardial Fibrosis on Cardiovascular Structure, Function and Functional Status in Heart Failure with Preserved Ejection Fraction. J Cardiovasc Transl Res. 2022 Dec;15(6):1436-1443. doi: 10.1007/s12265-022-10264-7. Epub 2022 Jul 5. PMID 35790651
- [Derived] Lewis GA, Rosala-Hallas A, Dodd S, Schelbert EB, Williams SG, Cunnington C, McDonagh T, Miller CA. Predictors of myocardial fibrosis and response to anti-fibrotic therapy in heart failure with preserved ejection fraction. Int J Cardiovasc Imaging. 2022 Jul;38(7):1569-1578. doi: 10.1007/s10554-022-02544-9. Epub 2022 Feb 9. PMID 35138474
- [Derived] Lewis GA, Dodd S, Clayton D, Bedson E, Eccleson H, Schelbert EB, Naish JH, Jimenez BD, Williams SG, Cunnington C, Ahmed FZ, Cooper A, Rajavarma Viswesvaraiah, Russell S, McDonagh T, Williamson PR, Miller CA. Pirfenidone in heart failure with preserved ejection fraction: a randomized phase 2 trial. Nat Med. 2021 Aug;27(8):1477-1482. doi: 10.1038/s41591-021-01452-0. Epub 2021 Aug 12. PMID 34385704
- [Derived] Lewis GA, Schelbert EB, Naish JH, Bedson E, Dodd S, Eccleson H, Clayton D, Jimenez BD, McDonagh T, Williams SG, Cooper A, Cunnington C, Ahmed FZ, Viswesvaraiah R, Russell S, Neubauer S, Williamson PR, Miller CA. Pirfenidone in Heart Failure with Preserved Ejection Fraction-Rationale and Design of the PIROUETTE Trial. Cardiovasc Drugs Ther. 2019 Aug;33(4):461-470. doi: 10.1007/s10557-019-06876-y. PMID 31069575